CLINICAL TRIAL: NCT06414369
Title: Effects of Diatermy in Patients With Fibromyalgia.
Acronym: FIBDIAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CamiloJDF
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; diathermy; pain; quality of life; chronic fatigue; anxiety
MeSH Terms: conditions — Fibromyalgia; Fever; Pain; Anxiety Disorders | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group will receive eight sessions of 20 minutes, for four weeks, twice a week.
  Interventions: Other: Diathermy
- Control group (Placebo Comparator): The treatment will be simulated during eight sessions of 20 minutes (machine will be off), for four weeks, twice a week.
  Interventions: Other: Simulated Diathermy

INTERVENTIONS:
Other: Diathermy — A DT equipment (CET 400 VA - RET 130 Watts - Winback, France), with a frequency of 500 kHz and intensity at 40% will be used. It will be applied utilizing a flat capacitive head 4 cm in diameter. It will be applied using longitudinal and transverse movements and a conductive cream for DT. DT will be used over the TP of the right and left trochanteric prominence. The settings will be calibrated so that patients fell no more than mild warmth during the treatment.
  Arms: Experimental group
Other: Simulated Diathermy — This same intervention that has been given to the experimental group, will be simulated as placebo in the control group; the DT will not be activated during administration.
  Arms: Control group

SUMMARY:
Diathermy is a non-invasive pain therapy based on the local application of high-frequency electromagnetic waves. This procedure produces deep heat promotes tissue repair and influences pain sensitivity. The main characteristic of fibromyalgia (FM) is generalized musculoskeletal pain. This may be accompanied by muscle and joint stiffness, sleep and mood disorders, anxiety and depression, cognitive dysfunction, and chronic fatigue. Endemic in developed countries, with a higher prevalence among women than men, and the etiology is still unknown. Diagnosis is made on chronic generalized pain and through the presence of tender points. The objective of this study will be to analyze the efficacy of diathermy on pain in patients with fibromyalgia

DETAILED DESCRIPTION:
The researchers aimed will be to observe the effect of diathermy (DT) on chronic fatigue, anxiety, and depression; analyze whether there are improvements in the impact of the disease in patients with FM after the application of DT; and check if there is an improvement in the quality of sleep after the application of DT.

The aim is to collect a sample of more than 30 patients with fibromyalgia. Variables to be collected include the overall pain experienced by the patients (Visual Analog Scale), Presure Pain Threshold using an algometer of the right and left trochanteric prominence, the Fibromyalgia Impact Questionnaire (FIQ) measures the impact of FM, the Hospital Anxiety and Depression Scale (HADS) to measure anxiety and depression, the Pittsburgh Sleep Quality Questionnaire (PSQI) to measure sleep quality and the modified Fatigue Impact Scale (MFI-S) to measure self-reported general fatigue.

Subjects will be randomized into two groups: a control group (CG) that will not recive treatment and a experimental group (EU).

ELIGIBILITY:
Inclusion Criteria:

* Experience chronic generalized pain and be diagnosed with FM for at least three months

Exclusion Criteria:

* Recent surgery, skin conditions unsuitable for DT application, presence of certain neuropathic conditions (lupus, rheumatoid arthritis, diabetic polyneuropathy), ongoing pharmacological treatment such as anticoagulants within three days before participation, any underlying medical conditions like fractures or tumors; cardiac pathologies including heart failure, uncontrolled arterial hypertension, arrhythmias, phlebitis thrombi arteriopathies; having a pacemaker or suffering from epilepsy.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pain (VAS) | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  visal analogue scale, on a scale of 1-10, with higher scores indicating more pain.
Pain (algometry) | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  Algometer, on a scale of 0-5. with higher scores indicating less pain.

SECONDARY OUTCOMES:
The impact of fibromyalgia. | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  The Fibromyalgia Impact Questionnaire (FIQ) measures the impact of FM. The values range between 0 and 100, with a higher score indicating a greater impact of the disease.
anxiety and depression | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  The Hospital Anxiety and Depression Scale (HADS) questionnaire, that consists of 14 items, divided into two subscales with 7 items each, using a Likert scale from 0 to 3. The odd-numbered items pertain to HADA, and the even-numbered ones relate to HADD. Each scale has a score range of 0-21 points. Higher scores indicate higher levels of anxiety and depression. Scores exceding 11 are classified as "cases," while those surpassing 8 are regarded as "probable cases" of anxiety and depression
sleep quality | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  The Pittsburgh Sleep Quality Questionnaire (PSQI)assesses seven dimensions: sleep quality, delay in falling asleep, duration of sleep, perceived effectiveness of sleep, disturbances during sleep, use of medication for sleeping, and daytime dysfunction. Each aspect is assigned a score from 0 to 3. Lower scores indicate no challenges in the specific areas while higher scores up to 3 indicate severe difficulties. The maximum achievable total score is 21 denoting critical sleep issues. A higher point total corresponds to a greater severity of sleep disorders.
self-reported general fatigue | base line; after finish the treatment (4 weeks) and 15 days after completing treatment.
  The modified Fatigue Impact Scale (MFI-S) with a a higher score that indicates a more severe condition.

CONTACTS AND LOCATIONS:
Overall Officials: Edurne Ú Docasar, Principal Investigator — University Camilo José Cela
Locations (1):
- University Camilo José Cela, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No